CLINICAL TRIAL: NCT03097731
Title: Epidemiological Screening of p.R101W and p.T179T IL10RA Mutation Rates in Henan Province, China
Brief Title: Epidemiological Screening of IL10RA Mutation Rate in China
Acronym: Yes
Status: Withdrawn | Type: Observational
Why Stopped: Preliminary tests found that some newborns heel blood amount could not meet the test needs.
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: 20170208
Record Dates: First submitted 2017-02-27; First posted 2017-03-31 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Digestive System Disease
Keywords: interleukin-10; inflammatory bowel disease
MeSH Terms: conditions — Digestive System Diseases; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Samples will be stored in 4 degrees refrigerator for the future research
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The presentation of IBD in early childhood is uncommon and the monogenetic defects, especially IL-10 signaling pathway play a key role in very early onset inflammatory bowel disease (VEO-IBD). IL-10 or IL-10R deficiency associated VEO-IBD is considered a rare disorder. To date, there were about 60 cases were reported all over the word. But in our Chinese VEO-IBD Collaboration Group, 42 patients with biallelic mutations affecting IL10R genes were identified from 93 VEO-IBD patients, and the mutation sites are highly concentrated, including 83.9% (26/31) with p.R101W and 55% p.T179T (17/31) mutation, and the proportion of patients from Henan( A province of China) is higher. So we speculate that IL-10RA mutation may not be very rare, and the frequency of heterozygote subjects might be higher than suspected.

DETAILED DESCRIPTION:
1. The mutation rates of p.R101W and p.T179T IL10RA in Henan newborn.
2. Is there any clinical symptoms in children with IL-10RA-deficient? and the onset of the symptoms.
3. Whether the intestinal permeability is normal in heterozygote subjects.

ELIGIBILITY:
Inclusion Criteria:

* In the study period, all newborns in the selected hospita

Exclusion Criteria:

* Children whose guardian refused to participate in the study

Ages: 24 Hours to 28 Days | Sex: All
Age Groups: Child
Study Population: In the study period, all newborns in the selected hospital were included.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-07-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
The mutation rate of IL-10RA in chinese | From birth to 3 years old
  All present mutations in IL-10RA

CONTACTS AND LOCATIONS:
Overall Officials: Ying Huang, MD and PhD, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's hospital of Fudan university, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided